CLINICAL TRIAL: NCT04709250
Title: Evaluating the Analgesic Efficacy of Combined Individual Nerve Block in Comparison to Interscalene Nerve Block in Patients Undergoing Shoulder Arthroscopic Assisted Adhesiolysis
Brief Title: Evaluating the Analgesic Efficacy of Combined Individual Nerve Block in Comparison to Interscalene Nerve Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rania Maher Hussien, MD, Assistant professor of Anaesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FMASU R 131/2020
Record Dates: First submitted 2021-01-07; First posted 2021-01-14 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A: receive ultrasound-guided interscalene block (Active Comparator): The patient will be put in the supine position, with the arm adducted a high-frequency linear ultrasound probe is oriented transversely across the lateral neck. When visualizing the ''stoplight sign,''15 to 30 mL of 0.25% bupivacaine consistent with the overall local anaesthetic dosing of less than 2.5 mg/kg. will be injected with low pressures to avoid intraneural injection.
  Interventions: Procedure: interscalene block; Drug: bupivacaine
- group B: receive ultrasound-guided selective nerve block (Active Comparator): The patient will be put in the sitting position, a linear 38-mm high frequency 10-12 MHz transducer will be placed first on the scapula to obtain a view of the suprascapular nerve a 22 G, 8 cm needle will be advanced in-plane and a total of 5-8 mL of 0.25% bupivacaine is injected then the arm adducted the linear probe will be placed at the junction of the pectoralis major muscle and the biceps muscle such that the axillary artery will be visualized in cross-section The probe will be moved towards the biceps muscle (laterally) until the musculocutaneous nerve is visualized and8 ml of 0.25% bupivacaine will be injected
  Interventions: Procedure: selective nerve block; Drug: bupivacaine

INTERVENTIONS:
Procedure: interscalene block — The patient will be put in the supine position, with the arm adducted a high-frequency linear ultrasound probe is oriented transversely across the lateral neck. When visualizing the ''stoplight sign,''15 to 30 mL of 0.25% bupivacaine will be injected
  Arms: group A: receive ultrasound-guided interscalene block
Procedure: selective nerve block — the patient will be put in the sitting position, linear 38-mm high frequency 10-12 MHz transducer will be placed first on the scapula to view of the suprascapular nerve. 5-8 mL of 0.25% bupivacaine is injected to block the SSN.
  The ultrasound probe put on the posterior aspect of the shoulder to view the circumflex artery, 10 mL of 0.25% bupivacaine this will lead to loss of sensation over the deltoid.lateral pectoral nerve block (LPNB) will be done by injecting a volume of 8 ml of a 0.25% bupivacaine The probe will be moved towards the biceps muscle until the musculocutaneous nerve is seen and 8 ml of 0.25% bupivacaine will be injected.
  Arms: group B: receive ultrasound-guided selective nerve block
Drug: bupivacaine — bupivacaine

SUMMARY:
Patients undergoing total shoulder arthroscopic adhesiolysis may experience severe postoperative pain. Inadequate pain management can result in unfavourable hospital outcomes and the development of persistent neuropathic manifestation the aim of the study is to compare both ultrasound techniques (combined individual nerve block to interscalene nerve block) as regards the postoperative analgesic effect and shoulder range of movement.

DETAILED DESCRIPTION:
60 patients will be attached to standard monitoring, will have a secured intravenous line Then the skin overlying the procedure area will be sterilized. all patients will be randomly divided into two equal groups; group A will receive ultrasound-guided interscalene block (ISNB), and group B will receive ultrasound-guided selective nerve block (SNB) of the following nerves; suprascapular nerve block (SSNB), axillary nerve block (ANB), lateral pectoral nerve block (LPNB) and musculocutaneous nerve block (MCNB).

after delivering the nerve block and confirming sensory blockade by loss of cold sensation, all the patients will receive general anaesthesia with endotracheal intubation using Propofol 200mg, Atracurium 0.5 mg/kg, 100 micrograms fentanyl.

After the procedure ends, the patient will be extubated and transferred to the postoperative anaesthesia care unit. All patients will receive patient-controlled analgesia (PCA) in the form ketorolac 30 mg and paracetamol one-gram iv infusion.

The following parameter will be assessed and measured;

1. Intra-operative inhalation agent consumption
2. Intraoperative opioid consumption (fentanyl) if required.
3. Duration of postoperative analgesia and time for first rescue analgesia will be recorded. Rescue analgesia in the form of 100mg pethidine IM and 1 gm paracetamol IV will be given on the first call for analgesia and then repeated on demand. The total dose of pethidine and paracetamol are given throughout the first 24 hours will be recorded.
4. The time for asking for rescue analgesia in the first 24 h and the dose of the analgesic used will also be recorded.
5. The degree of postoperative pain assessed by Visual Analogue Scale (VAS)
6. Duration of the block: time from completing LA injection till complete recovery of sensory function, i.e., the patient feels a cold sensation
7. Postoperative range of motion of the operated shoulder
8. Patients" satisfaction (yes or no or somewhat satisfied)
9. Block-related complications will be also recorded e.g. paraesthesia, and postoperative motor weakness 24 hours after the surgery, pneumothorax and vascular puncture.

ELIGIBILITY:
Inclusion Criteria:

* ASA I, II
* scheduled for arthroscopic assisted adhesiolysis

Exclusion Criteria:

* restrictive lung disease,
* refusal of the procedure,
* coagulopathy,
* allergy to any of the used medications

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
the duration of postoperative analgesia | 24 hours postoperative
  postoperative pain by visual analogue scale (VAS) a 10 point scale where 1 means no pain and 10 means worst pain ever

SECONDARY OUTCOMES:
range of motion of the operated shoulder | 24 hours postoperative
  free or limited

CONTACTS AND LOCATIONS:
Overall Officials: Fathy M Tash, MD, Study Chair — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt